CLINICAL TRIAL: NCT03242239
Title: A Randomized, Double-Blind, Parallel, Phase I Pharmacokinetic Trial Comparing The Potential Biosimilar ALT02(Trastuzumab) With Herceptin in Healthy Volunteers
Brief Title: A Comparing Study Between ALT02(Trastuzumab Biosimilar) and Herceptin® in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alteogen, Inc. (Industry)
Collaborators: Cristália Produtos Químicos Farmacêuticos Ltda. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALT02
Record Dates: First submitted 2017-08-02; First posted 2017-08-08 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Healthy
Keywords: HER2 Positive Breast Cancer; Trastuzumab; Biosimilar

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ALT02 (Experimental)
  Interventions: Biological: ALT02
- EU-licensed Herceptin (Active Comparator)
  Interventions: Biological: EU-licensed Herceptin
- US-licensed Herceptin (Active Comparator)
  Interventions: Biological: US-licensed Herceptin

INTERVENTIONS:
Biological: ALT02
  Arms: ALT02
Biological: EU-licensed Herceptin
  Arms: EU-licensed Herceptin
Biological: US-licensed Herceptin
  Arms: US-licensed Herceptin

SUMMARY:
The purpose of this study is to compare ALT02 (Trastuzumab biosimilar) and Herceptin® (US-licensed Trastuzumab and EU-licensed Trastuzumab) in healthy male subjects about the pharmacokinetics, safety, tolerability and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* Have a body weight over 50.0 kg and a body mass index over than 18.5 and less than 30.0 kg/m², inclusive.

Exclusion Criteria:

* Any clinically significant abnormality or abnormal laboratory test results found during medical screening or positive test for hepatitis B, hepatitis C, or HIV found during medical screening.
* Positive urine drug screen or alcohol breath test at screening.
* History of allergic reactions to trastuzumab, benzyl alcohol, murine proteins, or other related drugs.
* Any reason which, in the opinion of the Qualified Investigator, would prevent the subject from participating in the study.
* Clinically significant electrocardiogram (ECG) abnormalities or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
* History of significant alcohol abuse within one year prior to screening or regular use of alcohol within six months prior to the screening visit (more than fourteen units of alcohol per week [1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).
* History of significant drug abuse within one year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP], and crack) within 1 year prior to screening.
* Use of trastuzumab or another monoclonal antibody for a medical condition or in the context of another clinical trial.
* Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to dosing, administration of a biological product in the context of a clinical research study within 90 days prior to dosing, or concomitant participation in an investigational study involving no drug or device administration.
* Use of medication other than topical products without significant systemic absorption:

  1. prescription medication within 14 days prior to dose administration;
  2. over-the-counter products including natural health products (e.g. food supplements and herbal supplements) within 7 days prior to dosing, with the exception of the occasional use of acetaminophen (up to 2 g daily);
  3. a depot injection or an implant of any drug within 3 months prior to dose administration.
* Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to dosing.
* Hemoglobin <128 g/L and hematocrit <0.37 L/L at screening.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2016-02-09 (Actual); Primary Completion 2016-08-04 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
AUC0-inf: area under the concentration-time curve from time zero to infinity | 43 days

SECONDARY OUTCOMES:
AUC0-t: area under the concentration-time curve from time zero to the last non-zero concentration | 43 days
Cmax: maximum observed concentration | 43 days
Tmax: time of observed Cmax | 43 days
Kel: apparent terminal elimination rate constant | 43 days
T½ el: apparent terminal half-life | 43 days
CL: apparent body clearance, calculated as Dose/AUC0-inf | 43 days
Vd: apparent volume of distribution, calculated as Dose/(kel x AUC0-inf) | 43 days